CLINICAL TRIAL: NCT06139536
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BAT4706 Injection Combined With BAT1308 Injection in Patients With Advanced Solid Tumors
Brief Title: Assessment of Safety, Tolerability and Pharmacokinetics With BAT4706 and BAT1308 in Advanced Solid Tumors Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-4706-1308-001-CR
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A/ Standard 3+3 1.0mg/kg of BAT4706 with 300mg of BAT1308 (Experimental): Drug: BAT4706 injection, Dosage: 1.0mg/kg, Frequency: once every 3 weeks, Duration: 3 month.
  Drug: BAT1308 injection, Dosage: 300mg, Frequency: once every 3 weeks, Duration: 1 year.
  Interventions: Drug: BAT4706 Injection; Drug: BAT1308 Injection
- B/ Standard 3+3 2.0mg/kg of BAT4706 with 300mg of BAT1308 (Experimental): Drug: BAT4706 injection, Dosage: 2.0mg/kg, Frequency: once every 3 weeks, Duration: 3 month.
  Drug: BAT1308 injection, Dosage: 300mg, Frequency: once every 3 weeks, Duration: 1 year.
  Interventions: Drug: BAT4706 Injection; Drug: BAT1308 Injection
- C/ Standard 3+3 3.0mg/kg of BAT4706 with 300mg of BAT1308 (Experimental): Drug: BAT4706 injection, Dosage: 3.0mg/kg, Frequency: once every 3 weeks, Duration: 3 month.
  Drug: BAT1308 injection, Dosage: 300mg, Frequency: once every 3 weeks, Duration: 1 year.
  Interventions: Drug: BAT4706 Injection; Drug: BAT1308 Injection
- D/ Standard 3+3 6.0mg/kg of BAT4706 with 300mg of BAT1308 (Experimental): Drug: BAT4706 injection, Dosage: 6.0mg/kg, Frequency: once every 3 weeks, Duration: 3 month.
  Drug: BAT1308 injection, Dosage: 300mg, Frequency: once every 3 weeks, Duration: 1 year.
  Interventions: Drug: BAT4706 Injection; Drug: BAT1308 Injection
- E/ Standard 3+3 10.0mg/kg of BAT4706 with 300mg of BAT1308 (Experimental): Drug: BAT4706 injection, Dosage: 10mg/kg, Frequency: once every 3 weeks, Duration: 3 month.
  Drug: BAT1308 injection, Dosage: 300mg, Frequency: once every 3 weeks, Duration: 1 year.
  Interventions: Drug: BAT4706 Injection; Drug: BAT1308 Injection

INTERVENTIONS:
Drug: BAT4706 Injection — Intravenous infusion, 3 weeks one cycle(Q3W), Administer on the first day of each cycle. In the first four cycles, administration starting with BAT1308, and then administering BAT4706 on the same day. Maintain administration of BAT1308 monotherapy after four cycles.
  Other Names: Fc-glycosylated recombinant fully humanized anti-CTLA-4 monoclonal antibody injection
Drug: BAT1308 Injection — Intravenous infusion, 3 weeks one cycle(Q3W), Administer on the first day of each cycle. In the first four cycles, administration starting with BAT1308, and then administering BAT4706 on the same day. Maintain administration of BAT1308 monotherapy after four cycles.
  Other Names: Recombinant humanized anti PD-1 monoclonal antibody injection

SUMMARY:
This is a Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BAT4706 Injection Combined With BAT1308 Injection in Patients With Advanced Solid Tumors.

DETAILED DESCRIPTION:
The goal of this interventional study is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of BAT4706 injection combined with BAT1308 injection in patients with advanced solid tumors, explore the maximum tolerable dose. The study is generally divided into two stages. In the first stage, the "3+3" dose increasing rule is proposed to explore the safety and tolerability, subject will be given BAT1308 injection and BAT4706 injection through Intravenous infusion in the first four cycles, and then maintain administration of BAT1308 monotherapy after four cycles until 18 cycles; In the second stage, based on the preliminary safety and efficacy results of the previous stage, appropriate doses and tumor types were selected for extended research, in order to further explore the safety and clinical effectiveness of BAT4706 injection and BAT1308 injection in the combined administration mode.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent.
* Study population:

  1. Dose increasing stage:Patients with advanced malignant solid tumors who have been pathologically confirmed, have failed to standard treatment, or are intolerant to standard treatment.
  2. Dose expansion stage: Divided into 3 queues:

     1. Queue A: Patient with locally advanced or metastatic non-small cell lung cancer (NSCLC) confirmed by pathology, failed to standard treatment, or are intolerant to standard treatment. And it must meet the following requirements: a) Previous PD-L1 test results have been obtained; Or b) Provide previously stored tumor tissue samples or fresh biopsy tumor lesion tissue for PD-L1 testing at the site before the first medication use;
     2. Queue B: Advanced microsatellite stable (pMMR/MSS) colorectal cancer confirmed by pathology, with disease progression after receiving at least 2 standard chemotherapy regimens/lines, and no liver metastasis or resection/ablation liver metastasis.
     3. Queue C: Patient with Hepatocellular carcinoma confirmed by pathology, refractory to at least 1 line of previous systemic treatment, and intolerant to this treatment.
* An evaluable tumor focus was necessary in the dose escalation stage, and at least one measurable tumor focus in the dose expanding stage(according to RECIST 1.1 standard).
* ECOG should be 0-1 in the dose escalation stage, and be 0-2 in the dose expanding stage.
* The expected survival period is more than 12 weeks base on the evaluation of the investigator.
* Enough organs, bone marrow reserve function.
* Female patients with fertility must undergo a serum pregnancy test during the screening period, and the result is negative. Patient must agree to take effective contraceptive methods to prevent pregnancy.

Exclusion Criteria:

* Have received any other clinical trial treatment or participated in a medical device clinical study within 4 weeks prior to the first administration of the study drug.
* Previously failed to receive CTLA-4 monoclonal antibody treatment.
* Received other tumor treatments within 4 weeks prior to the first administration of the study drug, such as chemotherapy, radiotherapy (palliative radiotherapy must be completed within 2 weeks prior to the first administration), targeted therapy/immunotherapy (with a minimum interval of 4 weeks or at least 5 half-lives, whichever is shorter), hormone therapy (excluding alternative therapy).
* Prior to the first administration of the investigational drug, there were still cases of AE caused by previous anti-tumor therapy that were greater than level 1 (CTCAE5.0).
* Having undergone major surgery (such as craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first administration of the study drug, major surgery is defined as a level 3 or 4 surgery; Individuals with a history of organ transplant surgery.
* Primary central nervous system tumor or symptomatic central nervous system metastasis, meningeal metastasis, or previous history of epilepsy. Excluding patients with central nervous system metastasis who are clinically asymptomatic or have symptoms but have been judged stable by investigator.
* If other malignant tumors have been diagnosed within the past 5 years, or if previous malignant tumors have been cured for less than 5 years, the first pathological diagnosis shall prevail. Except radical skin basal cell carcinoma, skin squamous cell carcinoma or carcinoma in situ (such as breast cancer in situ, cervical carcinoma in situ).
* Severe cardiovascular disease: Heart failure with a New York Heart Association(NYHA) rating of 2 or above, left ventricular ejection fraction (LVEF) less than 50%, unstable arrhythmia or unstable angina, uncontrollable hypertension (defined in this protocol as systolic blood pressure>150mmHg and/or diastolic blood pressure>100mmHg after treatment, although the optimal antihypertensive treatment is used).
* Patients with a history of autoimmune diseases (those who undergo thyroid hormone replacement therapy to control stable hypothyroidism can be included in the group); Patients who are using immunosuppressive agents or systemic or absorbable local hormone therapy to achieve immunosuppressive effects (dosage>10mg/day of prednisone or other therapeutic hormones) and continue to use the study drug within 2 weeks before the first administration.
* Active infections with clinical significance that require intravenous antibiotics, including active pulmonary tuberculosis patients.
* Patients with uncontrolled or requiring drainage of pleural, pericardial, or abdominal effusion.
* Individuals at risk of thrombosis or bleeding.
* Individuals infected with the following diseases: human immunodeficiency virus (HIV) infection; Treponema pallidum antibody positive; Active hepatitis B virus infected; Hepatitis C virus infected.
* Received or planned to receive live/attenuated vaccines within 4 weeks prior to screening or during the study period.
* Known to have experienced severe hypersensitivity reactions to any monoclonal antibody.
* Patients who have a known history of abuse or drug use of psychotropic substances and are believed to affect compliance with this study.
* Pregnant or lactating women.
* The study participants who were considered unsuitable for the study by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | The first administration cycle(21 days)
  The following AEs related to the study drug occurred from day 1 to day 21 after administration in the first cycle:
  ≥grade 3 of non hematological toxicity (except for nausea, vomiting, and diarrhea that can be relieved within 3 days of supportive treatment, and those who recover within 2 hours of symptomatic treatment of infusion reactions); ≥grade 4 of Hematological toxicity(including ≥ 3 grade neutropenia with fever; however, grade 4 neutropenia requires a duration of ≥ 7 days to determine DLT);≥ grade 4 thrombocytopenia or grade 3 thrombocytopenia with bleeding.
Vital signs | Through study completion, 1 year
  Number of cases with abnormal vital signs results
Physical examination | Through study completion, 1 year
  Number of cases with abnormal physical examination results
Laboratory Examination | Through study completion, 1 year
  Number of cases with abnormal laboratory examination results
Electrocardiogram | Through study completion, 1 year
  Number of cases with abnormal electrocardiogram results
Echocardiography | Through study completion, 1 year
  Number of cases with abnormal echocardiography results
Adverse event | Through study completion, 1 year
  Number of cases with all adverse medical events that occur after the subject receives the investigational drug assessed by CTCAE V5.0

SECONDARY OUTCOMES:
Pharmacokinetic | Every cycle until 18 cycles (one cycle equals 3 weeks)
  Cmax
Immunogenicity | Every cycle until 18 cycles (one cycle equals 3 weeks)
  Presence of anti drug antibody (ADA)/Neutralizing antibodies (NAb)
Objective response rate (ORR) | Through study completion, 1 year
  Refer to the proportion of subjects defined as complete remission (CR) and partial remission (PR)
Best Overall Response Rate(BORR) | Through study completion, 1 year
  The proportion of subjects with complete response (CR) and partial response (PR) as the optimal ORR in tumor efficacy evaluation
Progression-Free Survival(PFS) | Through study completion, 1 year
  The time from the first administration to the occurrence of objective tumor progression or all cause death
Duration of Response(DOR) | Through study completion, 1 year
  DoR is defined as the time between the first assessment of objective remission of a tumor and death from any cause before the first assessment of Disease progression (PD) , reflecting the duration of ORR.
Overall Survival(OS) | Through study completion, 1 year
  The time from the date of first administration to the occurrence of death due to any cause. Subjects who were still alive at the time of analysis will use the date of their last contact as the deadline.

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital
Locations (3):
- China (3):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - Linyi Cancer Hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: No